CLINICAL TRIAL: NCT04396522
Title: Application of Serial Body Composition Change for Risk Prediction in Treating Patients With Severe Pneumonia
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900375B0
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Pneumonia
Keywords: pneumonia, sepsis, body composition
MeSH Terms: conditions — Pneumonia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: noninvasively Bio-electrical Impedance Analysis (BIA) — By means of noninvasively Bio-electrical Impedance Analysis (BIA) to measure body composition, which divides body weight into different components such as lean body mass and fat mass.

SUMMARY:
We hypothesize that serial changes of body composition in patients with pneumonia can help clinician to monitor prognosis. It was associated with underlying immune response.

DETAILED DESCRIPTION:
Specific aims:

1. Can serial body composition data be useful for predicting outcomes of patients with pneumonia? (developing sepsis, organ failure, admission to ICU, length of ICU, survival, length of stay in hospital, prolonged mechanical ventilation,..)
2. Can serial body composition data be integrated into both immune status alternatives (e.g., white blood cell (WBC) count, segment/monocyte ratio, pulse pressure) in such critical illness and monitoring responses (SOFA score, labs) for severe pneumonia patients?
3. Can serial body composition data reflect clinical variables in patients with pneumonia, and even altered by nutrition intake? (e.g., compare association between nutrition intake amount and groups stratified by body composition, blood pressure, nutritional intake, …)

ELIGIBILITY:
Inclusion Criteria:

Adult patients with pneumonia admitted to the thoracic ward or medical intensive care unit of Kaohsiung Chang Gung Memorial Hospital

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pneumonia admitted to the thoracic ward or medical intensive care unit of the Kaohsiung Chang Gung Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
ICU Days | During hospitalization， "through study completion, an average of 1 year"
  length of stay in ICU
Ventilation days | up to 24 weeks
  days of mechanical ventilation
sepsis free days | up to 24 weeks
  the cure day of sepsis
mortality | During hospitalization， "through study completion, an average of 1 year"
  death rate
Change in Total Body Water | Change from Baseline Total Body Water at day 8
  Change in Total Body Water
Change in Percentage of Body Fat | Change from Baseline Percentage of Body Fat at day 8
  Change in Percentage of Body Fat
Change in Soft Lean Mass | Change from Baseline Soft Lean Mass at day 8
  Change in Soft Lean Mass
Change in segment/monocyte ratio | Change from Baseline Segment count to monocyte count ratio at day 8
  Change in Segment count to monocyte count ratio

CONTACTS AND LOCATIONS:
Overall Officials: WEN-FENG Fang, Principal Investigator
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to disclose information about individual patients

REFERENCES:
- [Background] Wunderink RG, Waterer GW. Community-acquired pneumonia. N Engl J Med. 2014 May 8;370(19):1863. doi: 10.1056/NEJMc1402692. No abstract available. PMID 24806181
- [Background] Postma DF, van Werkhoven CH, van Elden LJ, Thijsen SF, Hoepelman AI, Kluytmans JA, Boersma WG, Compaijen CJ, van der Wall E, Prins JM, Oosterheert JJ, Bonten MJ; CAP-START Study Group. Antibiotic treatment strategies for community-acquired pneumonia in adults. N Engl J Med. 2015 Apr 2;372(14):1312-23. doi: 10.1056/NEJMoa1406330. PMID 25830421
- [Background] Fang WF, Yang KY, Wu CL, Yu CJ, Chen CW, Tu CY, Lin MC. Application and comparison of scoring indices to predict outcomes in patients with healthcare-associated pneumonia. Crit Care. 2011;15(1):R32. doi: 10.1186/cc9979. Epub 2011 Jan 19. PMID 21247444
- [Background] Fang WF, Douglas IS, Chen YM, Lin CY, Kao HC, Fang YT, Huang CH, Chang YT, Huang KT, Wang YH, Wang CC, Lin MC. Development and validation of immune dysfunction score to predict 28-day mortality of sepsis patients. PLoS One. 2017 Oct 26;12(10):e0187088. doi: 10.1371/journal.pone.0187088. eCollection 2017. PMID 29073262
- [Background] Tseng CC, Fang WF, Leung SY, Chen HC, Chang YC, Wang CC, Chang HC, Lin MC. Impact of serum biomarkers and clinical factors on intensive care unit mortality and 6-month outcome in relatively healthy patients with severe pneumonia and acute respiratory distress syndrome. Dis Markers. 2014;2014:804654. doi: 10.1155/2014/804654. Epub 2014 Mar 3. PMID 24723739
- [Background] Phua J, Koh Y, Du B, Tang YQ, Divatia JV, Tan CC, Gomersall CD, Faruq MO, Shrestha BR, Gia Binh N, Arabi YM, Salahuddin N, Wahyuprajitno B, Tu ML, Wahab AY, Hameed AA, Nishimura M, Procyshyn M, Chan YH; MOSAICS Study Group. Management of severe sepsis in patients admitted to Asian intensive care units: prospective cohort study. BMJ. 2011 Jun 13;342:d3245. doi: 10.1136/bmj.d3245. PMID 21669950
- [Background] Manga G, Calin GA, Manuc M, Droc G, Tudor S. New Definitions of Sepsis and the Quest for Specific Biomarkers. Are the miRNAs the Answer? Chirurgia (Bucur). 2018 Jul-Aug;113(4):464-468. doi: 10.21614/chirurgia.113.4.464. PMID 30183576
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Torres A, Niederman MS, Chastre J, Ewig S, Fernandez-Vandellos P, Hanberger H, Kollef M, Li Bassi G, Luna CM, Martin-Loeches I, Paiva JA, Read RC, Rigau D, Timsit JF, Welte T, Wunderink R. International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia: Guidelines for the management of hospital-acquired pneumonia (HAP)/ventilator-associated pneumonia (VAP) of the European Respiratory Society (ERS), European Society of Intensive Care Medicine (ESICM), European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and Asociacion Latinoamericana del Torax (ALAT). Eur Respir J. 2017 Sep 10;50(3):1700582. doi: 10.1183/13993003.00582-2017. Print 2017 Sep. PMID 28890434
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Fang WF, Chen YM, Lin CY, Huang KT, Kao HC, Fang YT, Huang CH, Chang YT, Wang YH, Wang CC, Lin MC. Immune profiles and clinical outcomes between sepsis patients with or without active cancer requiring admission to intensive care units. PLoS One. 2017 Jul 10;12(7):e0179749. doi: 10.1371/journal.pone.0179749. eCollection 2017. PMID 28692671
- [Background] Tseng CC, Fang WF, Huang KT, Chang PW, Tu ML, Shiang YP, Douglas IS, Lin MC. Risk factors for mortality in patients with nosocomial Stenotrophomonas maltophilia pneumonia. Infect Control Hosp Epidemiol. 2009 Dec;30(12):1193-202. doi: 10.1086/648455. PMID 19852664
- [Background] Chen YM, Fang WF, Kao HC, Chen HC, Tsai YC, Shen LS, Li CL, Chang HC, Huang KT, Lin MC, Wang CC, Chao TY. Influencing factors of successful eradication of multidrug-resistant Acinetobacter baumannii in the respiratory tract with aerosolized colistin. Biomed J. 2014 Sep-Oct;37(5):314-20. doi: 10.4103/2319-4170.132879. PMID 25179700
- [Background] Tseng CC, Liu SF, Wang CC, Tu ML, Chung YH, Lin MC, Fang WF. Impact of clinical severity index, infective pathogens, and initial empiric antibiotic use on hospital mortality in patients with ventilator-associated pneumonia. Am J Infect Control. 2012 Sep;40(7):648-52. doi: 10.1016/j.ajic.2011.08.017. Epub 2012 Jan 13. PMID 22243991
- [Background] Huang KT, Tseng CC, Fang WF, Lin MC. An early predictor of the outcome of patients with ventilator-associated pneumonia. Chang Gung Med J. 2010 May-Jun;33(3):274-82. PMID 20584505
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Berman SJ, Johnson EW, Nakatsu C, Alkan M, Chen R, LeDuc J. Burden of infection in patients with end-stage renal disease requiring long-term dialysis. Clin Infect Dis. 2004 Dec 15;39(12):1747-53. doi: 10.1086/424516. Epub 2004 Nov 18. PMID 15578394
- [Background] Lee JH, Moon JC. Clinical characteristics of patients with hemodialysis-associated pneumonia compared to patients with non-hemodialysis community-onset pneumonia. Respir Med. 2016 Feb;111:84-90. doi: 10.1016/j.rmed.2015.12.009. Epub 2015 Dec 25. PMID 26777263
- [Background] Lim CW, Choi Y, An CH, Park SJ, Hwang HJ, Chung JH, Min JW. Facility characteristics as independent prognostic factors of nursing home-acquired pneumonia. Korean J Intern Med. 2016 Mar;31(2):296-304. doi: 10.3904/kjim.2014.256. Epub 2016 Feb 2. PMID 26837007
- [Background] Dhawan N, Pandya N, Khalili M, Bautista M, Duggal A, Bahl J, Gupta V. Predictors of mortality for nursing home-acquired pneumonia: a systematic review. Biomed Res Int. 2015;2015:285983. doi: 10.1155/2015/285983. Epub 2015 Mar 2. PMID 25821793
- [Background] Kao HC, Lai TY, Hung HL, Chen YM, Chou PA, Wang CC, Lin MC, Fang WF. Sequential oxygenation index and organ dysfunction assessment within the first 3 days of mechanical ventilation predict the outcome of adult patients with severe acute respiratory failure. ScientificWorldJournal. 2013;2013:413216. doi: 10.1155/2013/413216. Epub 2013 Feb 18. PMID 23476133
- [Background] Chang YC, Huang KT, Chen YM, Wang CC, Wang YH, Tseng CC, Lin MC, Fang WF. Ventilator Dependence Risk Score for the Prediction of Prolonged Mechanical Ventilation in Patients Who Survive Sepsis/Septic Shock with Respiratory Failure. Sci Rep. 2018 Apr 4;8(1):5650. doi: 10.1038/s41598-018-24028-4. PMID 29618837
- [Background] Hung KY, Chen YM, Wang CC, Wang YH, Lin CY, Chang YT, Huang KT, Lin MC, Fang WF. Insufficient Nutrition and Mortality Risk in Septic Patients Admitted to ICU with a Focus on Immune Dysfunction. Nutrients. 2019 Feb 10;11(2):367. doi: 10.3390/nu11020367. PMID 30744171
- [Background] Lin MC, Leung SY, Fang WF, Chin CH, Chung KF. Down-regulation of insulin-like growth factor I (IGF-I) in the mouse diaphragm during sepsis. Chang Gung Med J. 2010 Sep-Oct;33(5):501-8. PMID 20979700
- [Background] Chao WC, Tseng CH, Chien YC, Sheu CC, Tsai MJ, Fang WF, Chen YM, Kao KC, Hu HC, Perng WC, Yang KY, Chen WC, Liang SJ, Wu CL, Wang HC, Chan MC; TSIRC (Taiwan Severe Influenza Research Consortium). Association of day 4 cumulative fluid balance with mortality in critically ill patients with influenza: A multicenter retrospective cohort study in Taiwan. PLoS One. 2018 Jan 9;13(1):e0190952. doi: 10.1371/journal.pone.0190952. eCollection 2018. PMID 29315320
- [Background] Falagas ME, Kompoti M. Obesity and infection. Lancet Infect Dis. 2006 Jul;6(7):438-46. doi: 10.1016/S1473-3099(06)70523-0. PMID 16790384
- [Background] Hegde V, Dhurandhar NV. Microbes and obesity--interrelationship between infection, adipose tissue and the immune system. Clin Microbiol Infect. 2013 Apr;19(4):314-20. doi: 10.1111/1469-0691.12157. PMID 23506525
- [Background] Corrales-Medina VF, Valayam J, Serpa JA, Rueda AM, Musher DM. The obesity paradox in community-acquired bacterial pneumonia. Int J Infect Dis. 2011 Jan;15(1):e54-7. doi: 10.1016/j.ijid.2010.09.011. Epub 2010 Nov 20. PMID 21095152
- [Background] Arabi YM, Dara SI, Tamim HM, Rishu AH, Bouchama A, Khedr MK, Feinstein D, Parrillo JE, Wood KE, Keenan SP, Zanotti S, Martinka G, Kumar A, Kumar A; Cooperative Antimicrobial Therapy of Septic Shock (CATSS) Database Research Group. Clinical characteristics, sepsis interventions and outcomes in the obese patients with septic shock: an international multicenter cohort study. Crit Care. 2013 Apr 17;17(2):R72. doi: 10.1186/cc12680. PMID 23594407
- [Background] Maeda K, Akagi J. Muscle Mass Loss Is a Potential Predictor of 90-Day Mortality in Older Adults with Aspiration Pneumonia. J Am Geriatr Soc. 2017 Jan;65(1):e18-e22. doi: 10.1111/jgs.14543. Epub 2016 Nov 17. PMID 27858956
- [Background] Hung KY, Chiou TT, Wu CH, Liao YC, Chen CN, Yang PH, Wang HJ, Lee CT. Effects of Diet Intervention on Body Composition in the Elderly with Chronic Kidney Disease. Int J Med Sci. 2017 Jul 18;14(8):735-740. doi: 10.7150/ijms.19816. eCollection 2017. PMID 28824308
- [Background] Ischaki E, Papatheodorou G, Gaki E, Papa I, Koulouris N, Loukides S. Body mass and fat-free mass indices in COPD: relation with variables expressing disease severity. Chest. 2007 Jul;132(1):164-9. doi: 10.1378/chest.06-2789. Epub 2007 May 15. PMID 17505043
- [Background] Tamashiro KL, Hegeman MA, Nguyen MM, Melhorn SJ, Ma LY, Woods SC, Sakai RR. Dynamic body weight and body composition changes in response to subordination stress. Physiol Behav. 2007 Jul 24;91(4):440-8. doi: 10.1016/j.physbeh.2007.04.004. Epub 2007 Apr 12. PMID 17512562
- [Background] Reid CL, Murgatroyd PR, Wright A, Menon DK. Quantification of lean and fat tissue repletion following critical illness: a case report. Crit Care. 2008;12(3):R79. doi: 10.1186/cc6929. Epub 2008 Jun 17. PMID 18559097
- [Background] Lin TY, Peng CH, Hung SC, Tarng DC. Body composition is associated with clinical outcomes in patients with non-dialysis-dependent chronic kidney disease. Kidney Int. 2018 Mar;93(3):733-740. doi: 10.1016/j.kint.2017.08.025. PMID 29102374
- [Background] De Backer D, Dorman T. Surviving Sepsis Guidelines: A Continuous Move Toward Better Care of Patients With Sepsis. JAMA. 2017 Feb 28;317(8):807-808. doi: 10.1001/jama.2017.0059. No abstract available. PMID 28114630
- [Background] Feng JY, Fang WF, Wu CL, Yu CJ, Lin MC, Ku SC, Chen YC, Chen CW, Tu CY, Su WJ, Yang KY. Concomitant pulmonary tuberculosis in hospitalized healthcare-associated pneumonia in a tuberculosis endemic area: a multi-center retrospective study. PLoS One. 2012;7(5):e36832. doi: 10.1371/journal.pone.0036832. Epub 2012 May 22. PMID 22629334
- [Background] Arens C, Bajwa SA, Koch C, Siegler BH, Schneck E, Hecker A, Weiterer S, Lichtenstern C, Weigand MA, Uhle F. Sepsis-induced long-term immune paralysis--results of a descriptive, explorative study. Crit Care. 2016 Feb 29;20:93. doi: 10.1186/s13054-016-1233-5. PMID 27056672
- [Background] WF Fang CH, CY Lin, YT Fang, KT Huang, HC Kao, YH Wang, YT Chang, CC Wang, MC Lin. Immune Status and SeMo Score Predict Outcomes in Patients with Severe Sepsis. Am J Respir Crit Care Med. 2017;195:A1821.
- [Background] KY Hung WF, CH Huang, YM Chen, CY Lin, YT Chang, KT Huang, YH Wang, CC Wang, MC Lin. Body mass index (BMI) can help predict immune status and short-term survival in patients with sepsis admitted to ICU. Respirology (Carlton, Vic.). 2018;23(s2):AP460.
- [Background] WF Fang KH, YM Chen, YC Chong, YT Fang, KT Huang, YH Wang, H Yeh, YT Chang, CC Wang, MC Lin. Incremental Pulse Pressure Predicts Better Short-Term Outcomes in Patients with Sepsis Admitted to ICU. Am J Respir Crit Care Med. 2018;197:A6012.
- [Background] Lin FM, Feng JY, Fang WF, Wu CL, Yu CJ, Lin MC, Ku SC, Chen CW, Tu CY, Yang KY. Impact of prior pulmonary tuberculosis in treatment outcomes of HCAP and CAP patients in intensive care units. J Microbiol Immunol Infect. 2019 Apr;52(2):320-328. doi: 10.1016/j.jmii.2018.08.012. Epub 2018 Sep 5. PMID 30245205